CLINICAL TRIAL: NCT01508156
Title: A Phase I/IIa Study Assessing Single and Multiple Doses of HCV NS5A Inhibitor IDX719 in Healthy and HCV-Infected Subjects
Brief Title: Study of Hepatitis C Virus (HCV) Nonstructural Protein 5a (NS5A) Inhibitor IDX719 in Healthy and HCV-Infected Participants (MK-1894-001)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1894-001; IDX-06A-001 (Other: Idenix Pharmaceuticals, Inc)
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; treatment-naive
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — samatasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Healthy Participants (Experimental): Healthy participants take IDX719 (5 mg - 100 mg) or matching placebo by mouth as either 1 single dose or as 7 daily doses.
  Interventions: Drug: IDX719; Drug: Placebo
- Group B: HCV Participants (Experimental): Treatment-naive participants infected with HCV genotype (GT) 1, GT2, or GT3 take IDX719 (1 mg - 100 mg) or matching placebo as either 1 single dose or as 7 daily doses.
  Interventions: Drug: IDX719; Drug: Placebo

INTERVENTIONS:
Drug: IDX719 — IDX719 liquid suspension (1 - 100 mg) taken by mouth.
Drug: Placebo — Placebo liquid suspension matching IDX719 taken by mouth.

SUMMARY:
The purpose of the study is to test the safety and tolerability of different doses of IDX719 to find the best dose for future studies. The study will also assess the pharmacokinetics of IDX719. No formal hypotheses will be tested.

ELIGIBILITY:
Inclusion Criteria:

* All Participants
* Is in good general health.
* Agrees to use double-barrier method of birth control for at least 90 days after the last dose of study drugs.
* HCV Participants
* Has documented GT1, GT2, or GT3 chronic HCV infection.

Exclusion Criteria:

* All Participants
* Is pregnant or breastfeeding.

HCV Participants

* Has received prior HCV treatment.
* Is co-infected with hepatitis B virus (HBV) and/or human immunodeficiency virus (HIV).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants experiencing an adverse event (AE) | Up to 14 days
Percentage of participants experiencing serious AEs (SAEs) | Up to 14 days
Change in HCV ribonucleic acid (RNA) | Baseline and Day 10
Maximum plasma drug concentration (Cmax) | Pre-dose Day 1 to Day 13
Time to maximum plasma drug concentration (Tmax) | Pre-dose Day 1 to Day 13
Area under the plasma drug concentration-time curve (AUC) from time zero to time of last measurable concentration (AUC0-t) | Pre-dose Day 1 to Day 13
AUC from time zero to time 24 hours (AUC0-24h) | Pre-dose Day 1 to Day 1
AUC from time zero to time infinity (AUC0-~) | Pre-dose Day 1 to Day 13
Pre-dose trough plasma drug concentration (Ctrough) | Pre-dose Day 1
Observed terminal plasma drug concentration half-life (t1/2) | Pre-dose Day 1 to Day 13
Apparent oral total plasma drug clearance (CL/F) as Dose/AUC0-~ (single dose) or Dose/AUC0-t (multiple doses) | Pre-dose Day 1 to Day 13
Apparent oral total volume of distribution (Vz/F) | Pre-dose Day 1 to Day 13
Amount excreted in urine in each collection interval (Au) | Pre-dose Day 1 to Day 14
Cumulative urine excretion (Au0-t) | Pre-dose Day 1 to Day 14
Percentage of dose excreted in urine (% Dose excr) | Pre-dose Day 1 to Day 14
Renal clearance (CLr) | Pre-dose Day 1 to Day 14
Percentage of participants experiencing dose-limiting toxicity | Up to 8 days
Percentage of participants experiencing graded laboratory abnormalities | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Vince B, Hill JM, Lawitz EJ, O'Riordan W, Webster LR, Gruener DM, Mofsen RS, Murillo A, Donovan E, Chen J, McCarville JF, Sullivan-Bolyai JZ, Mayers D, Zhou XJ. A randomized, double-blind, multiple-dose study of the pan-genotypic NS5A inhibitor samatasvir in patients infected with hepatitis C virus genotype 1, 2, 3 or 4. J Hepatol. 2014 May;60(5):920-7. doi: 10.1016/j.jhep.2014.01.003. Epub 2014 Jan 14. PMID 24434503